CLINICAL TRIAL: NCT03668483
Title: Relation Between Upper and Lower Limb Muscle Strength With Exercise Capacity and Dyspnea in Patients With Awaiting Lung Transplantation
Brief Title: Relation Between Muscle Strength With Exercise Capacity and Dyspnea in LTx
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, esra pehlivan, Principal investigator, Istanbul Medipol University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Tx_Muscle strenght
Record Dates: First submitted 2018-09-11; First posted 2018-09-12 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2018-10

CONDITIONS: Lung Transplantation; Pulmonary Rehabilitation
Keywords: rehabilitation; exercise; maximal inspiratory pressure; walk test; muscle strength; dyspnea; lung transplantation
MeSH Terms: conditions — Motor Activity; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pulmonary Rehabilitation (Experimental): A 6-min walk test, peripheral and respiratory muscle strength measurements, and a dyspnea rating scale Mmrc will be applied to the lung transplantation candidates who are trained in 3-month hospital-based preoperative exercise training in the Pulmonary Rehabilitation unit. The tests will be carried out at the beginning and end of rehabilitation.
  Interventions: Other: Pulmonary rehabilitation

INTERVENTIONS:
Other: Pulmonary rehabilitation — A 6-min walk test, peripheral and respiratory muscle strength measurements, and a dyspnea rating scale Mmrc will be applied to the lung transplantation candidates who are trained in 3-month hospital-based preoperative exercise training in the Pulmonary Rehabilitation unit. The tests will be carried out at the beginning and end of rehabilitation.

SUMMARY:
Severe exercise intolerance and shortness of breath are present in lung transplant candidates. Clinical features that reveal these symptoms in terminal period lung patients vary and are unclear. The effect of peripheral muscle strength on exercise capacity and dyspnea will be examined in our study.

DETAILED DESCRIPTION:
Yedikule Chest Diseases Patients who have been accepted to participate in the pre-operative rehabilitation program at the Pulmonary Rehabilitation Unit will be included in the study. A 6-min walk test, peripheral and respiratory muscle strength measurements, and a dyspnea rating scale Mmrc will be applied to the lung transplantation candidates who are trained in 3-month hospital-based preoperative exercise training in the Pulmonary Rehabilitation unit. The tests will be carried out at the beginning and end of rehabilitation. At each testing session, the tests will be performed by the same physiotherapist. The correlations of the test data with each other will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* have a diagnosis of terminally severe lung disease,
* being listed for lung transplantation,
* medically stable,
* had no orthopedic or cardiac problems that would prevent them from exercising
* had no transfer problem to the pulmonary rehabilitation center.

Exclusion Criteria:

* Dont except to participate the study
* incompatibility with exhaust
* not completing the program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2018-09-20 (Actual); Primary Completion 2019-08-01 (Actual); Study Completion 2019-08-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline the muscle strength | 15 minutes
  Muscle strength will measure using a digital dynamometer (J-Tech Commander muscle testing device), wth three measurements make. Best result will be taken.
Changes from baseline the hand grip strength. | 5 minutes
  It was measured with hydraulic hand dynamometer calibrated in lbs.
Changes from baseline the maximum inspiratory muscle pressure | 15 minutes
  The mouth pressure measurement was performed with the Micro-RPM® instrument from SensorMEDIC. Patient placed a rubber mouthpiece with flanges, on the device, sealed their lips firmly around the mouthpiece, exhaled/inhaled slowly and completely, and then tried to breath in as hard as possible. The patient was allowed to rest for about a minute and the maneuver was repeated five times. Verbal or visual feedback was provided after each maneuver. The aim is that the variability between measurements is less than 10 cm H2O. The maximum value was obtained.
Changes from baseline the distance covered in six-minute walk test | 20 minutes
  The test was conducted in a 30-meter corridor in line with American Thoracic Society (ATS) guidelines. Patients were told that they should walk as fast as they can walk. Before and after the test, oxygen saturation, heart rate, Borg fatigue rating, and walking distance were recorded.
Changes from baseline the modified Medical Research Council (mMRC) scale | 5 minutes
  The mMRC Dyspnea Scale is best used to establish baseline functional impairment due to dyspnea attributable to respiratory disease; tracking the mMRC over time or with therapeutic interventions is of less certain clinical utility.The severity of dyspnea is rated on a scale of 0 to 4. "O" means no dyspnea perception, "4" means severe dyspnea perception.

CONTACTS AND LOCATIONS:
Locations (1):
- Yedikule Chest Disease Hospital, Istanbul, Zeytinburnu, Turkey (Türkiye)